CLINICAL TRIAL: NCT05157919
Title: Evaluation of a Mobile App to Promote Family Caregiver Engagement in Symptom Assessment and Management During Mechanical Ventilation in the Intensive Care Unit
Brief Title: Mobile App to Promote Family Caregiver Engagement in the Intensive Care Unit
Acronym: ICU-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 0625-17-EP
Record Dates: First submitted 2021-07-16; First posted 2021-12-15 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Family; Critical Care; Mobile Applications
Keywords: Caregiver; Critical Illness; Family; Psychological Distress; Family-Centered Nursing
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care continues. The caregiver will not get to use the app. The caregiver will be asked daily measures and the patient will be asked about thirst and anxiety daily when the patient is awake enough to answer these questions. The caregiver will be asked questions at 3 different times: Day 1, 24-48 hours after enrollment, and 2-4 weeks after the patient is discharged from the ICU.
- Intervention with App (Experimental): The caregiver gets access to use the app. Each day, investigators will ask the patient to rate their thirst and anxiety and the caregiver to answer daily measures through the application. The caregiver will be asked questions at 3 different times: Day 1, 24-48 hours after enrollment, and 2-4 weeks after the patient is discharged from the ICU. The caregiver will be taught how to use the app. The caregiver will be given the supplies that the caregiver needs to perform the symptom management intervention. Investigators will ask the caregiver to use the app at least once a day, but the caregiver can use it as much as desired while the patient is in the ICU.
  Interventions: Behavioral: ICU-Care

INTERVENTIONS:
Behavioral: ICU-Care — The mobile app intervention, ICU-CARE, will consist of 3 separate education modules, each approximately 5-7 minutes in length: (Module #1) ICU orientation, (Module #2) Symptom Assessment, (Module #3) Symptom Management
  Arms: Intervention with App

SUMMARY:
The purpose of this randomized controlled pilot trial is to develop and test mobile app, Intensive Care Unit-Caregiver Activation Response, and Engagement (ICU-CARE). ICU-CARE provides a simulated learning environment to encourage family caregivers of mechanically ventilated patients to assess two patient symptoms, thirst and anxiety, and perform specific nonpharmacologic comfort measures to help alleviate patient symptom burden.

DETAILED DESCRIPTION:
Critical care guidelines call for the liberal inclusion of family caregivers into bedside care, but despite convincing evidence that active family participation improves the patient and family experience as well as safety, quality, and delivery of care, critical care nurses have few evidence-based strategies to engage family caregivers as active participants in the provision of care in the intensive care unit (ICU). The broad objective of this proposal is to develop and test a mobile app, Intensive Care Unit-Caregiver Activation Response and Engagement [ICU-CARE]. ICU-CARE provides a simulated learning environment that incorporates established motivational learning theories to encourage family caregivers of mechanically ventilated patients to assess two patient symptoms, thirst and anxiety, and perform specific nonpharmacologic symptom management techniques to help alleviate the patient's symptom burden. This project, guided by the Individual and Family Self-Management Theory, aims to (1) Establish the feasibility and acceptability of the ICU-CARE intervention for family caregivers enrolled in the experimental arm; and (2) Determine the influence of the ICU-CARE intervention on the caregiver process characteristics, proximal caregiving outcomes, and distal caregiving outcomes as compared to family caregivers enrolled in the control arm. To address these study aims, a convenience sample of 60 family caregivers of mechanically ventilated patients will be recruited into this randomized controlled pilot trial. 30 participants will be enrolled to the control group which will receive usual care with routine caregiver support practices. Intervention participants (n=30) will be enrolled to an experimental condition ICU-CARE, that will consist of a theoretically grounded mobile app program to promote caregiver engagement in symptom assessment and management in the ICU. This project will help further define the scope, extent, and nature of patient and family engagement in the ICU, and if proven feasible, our intervention holds the potential to shift the ICU nursing practice paradigm by integrating family caregivers as dynamic partners in ICU care.

ELIGIBILITY:
Inclusion Criteria:

Adult Caregivers of mechanically ventilated ICU patients who are:

* Age 19 or older
* Able to understand English
* Able and willing to use the hospital-provided tablet devices
* Can view images on a screen and hear audio through a standard headset
* Have basic reading skills and the ability to read aloud

Critically ill patients in the ICU who are:

* Age 19 or older
* Mechanically ventilated
* Expected to require> 72 consecutive hours of mechanical ventilation during their ICU stay
* Calm, cooperative (a Richmond Agitation-Sedation Scale score between -5 and +1)
* Able to reliably report symptoms of thirst and anxiety per nursing assessment
* Have no documented hearing deficits
* Have a designated caregiver who visits frequently (daily for a minimum of 1 hour)

Exclusion Criteria:

Adult Caregivers of mechanically ventilated ICU patients who are:

* Caregivers of patients who are not currently undergoing mechanical ventilation
* Caregivers of patients who are not calm, cooperative (a Richmond Agitation- - Sedation Scale score between +2 and +4),
* Caregivers of patients who cannot reliably report symptoms of thirst and anxiety
* Caregivers of patients who have a documented hearing deficit.
* Caregivers who do not visit the patient frequently (at least once per day for a minimum of 1 hour as described by nursing staff)

Critically ill patients in the ICU who are:

* Recovering from any of the following surgeries: Glossectomy, Maxillectomy, Neck Dissection, Facial/neck flap
* Receiving aggressive ventilator support such as positive end expiratory pressure> 15cm of water, prone ventilation
* Not alert per nursing assessment (Richmond Agitation-Sedation Scale Score +2 or greater)
* Severe cognition or communication problems (i.e. coma as the main reason for intubation, dementia, severe delirium)
* Deafness

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Enrollment Feasibility of ICU-CARE | Through study completion, estimated 3 years.
  Total subjects screened, approached, consented and refused
Sustainability of ICU-CARE enrollment | Through study completion, estimated 3 years.
  Differential attrition rates - the number of subjects in each group that complete all study follow-up measures
Dosage of ICU-CARE | Through study completion, estimated 3 years.
  Number of doses of the intervention per participant
Acceptability of ICU-CARE | Through study completion, estimated 3 years.
  Total score of a modified version of the Educational Material Acceptability Instrument. Minimum Score = 11; Maximum Score = 55. Higher score indicates greater acceptance.

SECONDARY OUTCOMES:
Influence of ICU-CARE on Caregiver Process Characteristics - Caregiver Activation | At study enrollment, 24-48 hours after study enrollment, and 2-4 weeks after ICU discharge
  Caregiver activation as measured by Patient Activation Measure for Family Caregivers (CG-PAM). Minimum score = 1; Maximum Score = 4. Higher score indicates greater activation.
Influence of ICU-CARE on Caregiver Process Characteristics - Caregiver Self-efficacy | At study enrollment, 24-48 hours after study enrollment, and 2-4 weeks after ICU discharge
  Caregiver self-efficacy as measured by the Caregiver Self-Efficacy Scale (CaSES). Scale contains four sub-scales that are scored separately. Minimum Score =1; Maximal Score = 5. Higher scores indicate greater self-efficacy.
Influence of ICU-CARE on Caregiver Process Characteristics - Caregiver Preparedness | At study enrollment, 24-48 hours after study enrollment, and 2-4 weeks after ICU discharge
  Caregiver Preparedness as measured by the Preparedness for Caregiving Scale (Prep Scale). Minimum score = 0; Maximum score = 32. The higher the score the more prepared the caregiver feels for caregiving.
Influence of ICU-CARE on Proximal Caregiving Outcomes - Symptom Assessment | Once every 24 hours from the date the patient is enrolled in the trial to the date the patient is discharged from the ICU, an average of 2 weeks.
  Rate of symptom assessment behaviors - the number of times in a 24 hour period that the subject records a patient symptom assessment in the ICU-CARE app
Influence of ICU-CARE on Proximal Caregiving Outcomes - Symptom Management | Once every 24 hours from the date the patient is enrolled in the trial to the date the patient is discharged from the ICU, an average of 2 weeks.
  Rate of symptom management behaviors - the number of times in a 24 hour period that the subject records a patient symptom management technique in the ICU-CARE app
Influence of ICU-CARE on Proximal Caregiving Outcomes - Caregiver Anxiety | Once every 24 hours from the date the patient is enrolled in the trial to the date the patient is discharged from the ICU, an average of 2 weeks.
  Caregiver anxiety as measured by the State-Trait Anxiety Inventory (STAI-State). Minimum score = 0; Maximum score = 6. Higher scores indicate greater anxiety.
Influence of ICU-CARE on Proximal Caregiving Outcomes - Patient Thirst | Once every 24 hours from the date the patient is enrolled in the trial to the date the patient is discharged from the ICU, an average of 2 weeks.
  Patient thirst as measured by a 0-100 visual analogue scale for thirst (VAS-Thirst)
Influence of ICU-CARE on Proximal Caregiving Outcomes - Patient Anxiety | Once every 24 hours from the date the patient is enrolled in the trial to the date the patient is discharged from the ICU, an average of 2 weeks.
  Patient anxiety as measured by a 0-100 visual analogue scale for anxiety (VAS-Anxiety)
Influence of ICU-CARE on Distal Caregiving Outcomes - Caregiver Global Health Status | At study enrollment and 2-4 weeks after ICU discharge
  Caregiver Global Health Status as measured by the Patient-Reported Outcome Measure (PROMIS-10). 5 questions each on 2 (1-5) subscales (Global Physical Health, Global Mental Health). Once every 24 hours from the date the patient is enrolled in the trial to the date the patient is discharged from the ICU, an average of 2 weeks. Higher scores indicate a healthier patient.
Influence of ICU-CARE on Distal Caregiving Outcomes - Caregiver Anxiety & Depressive Symptoms | At study enrollment and 2-4 weeks after ICU discharge
  Caregiver anxiety and depressive symptoms as measured by the Hospital Anxiety and Depression Scale (HADS). Two sub-scales (Anxiety & Depression) scored separately. Minimum Score = 0; Maximum Score = 21. Higher score = higher anxiety and/or depression.
Influence of ICU-CARE on Distal Caregiving Outcomes - Caregiver Satisfaction | At study enrollment and 2-4 weeks after ICU discharge
  Caregiver satisfaction as measured by the Critical Care Family Satisfaction Survey (CCFSS). Minimum Score = 5; Maximum score = 25. Higher scores indicate greater satisfaction.
Influence of ICU-CARE on Distal Caregiving Outcomes - Caregiver ICU Experience | At study enrollment and 2-4 weeks after ICU discharge
  Overall impact of ICU experience for caregivers as measured by the Impact of Events Scale-Revised. Minimum Score = 0; Maximum Score = 88. Higher score indicates great impact of life event.
Influence of ICU-CARE on Distal Caregiving Outcomes - Patient Agitation | Once every 24 hours from the date the patient is enrolled in the trial to the date the patient is discharged from the ICU, an average of 2 weeks.
  Nurse documentation of patient agitation in the electronic health record
Influence of ICU-CARE on Distal Caregiving Outcomes - Patient Pain | Once every 24 hours from the date the patient is enrolled in the trial to the date the patient is discharged from the ICU, an average of 2 weeks.
  Nurse documentation of patient pain in the electronic health record
Influence of ICU-CARE on Distal Caregiving Outcomes - Duration of Ventilation | Once every 24 hours from the date the patient is enrolled in the trial to the date the patient is discharged from the ICU, an average of 2 weeks.
  Duration of mechanical ventilation
Influence of ICU-CARE on Distal Caregiving Outcomes - Sedative Exposure | Through study completion, estimated 3 years.
  Sedative exposure (sedation intensity and sedation frequency)

CONTACTS AND LOCATIONS:
Overall Officials: Breanna D Hetland, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Nebraska Medicine, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No